CLINICAL TRIAL: NCT04496557
Title: Feasibility Open Label Study Evaluating The Use Of Process-Instructed Self Neuro-Modulation (PRISM) For Post-Traumatic Stress Disorder
Acronym: PRISM
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The investigators received funding for a near-identical FDA regulated trial before opening this study to enrollment - the IRB requested closure of the unfunded pilot trial to create a new submission.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20-00792
Record Dates: First submitted 2020-07-29; First posted 2020-08-03 (Actual); Last update posted 2021-06-14 (Actual); Status verified 2021-06

CONDITIONS: Post-traumatic Stress Disorder
MeSH Terms: conditions — Stress Disorders, Post-Traumatic

STUDY DESIGN:
Intervention Model Description: single-arm, open-label feasibility study
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Patients diagnosed with PTSD (Experimental): 7-15 men and women with PTSD will be recruited from the community and from local clinical programs through a multi-modal outreach program.
  Interventions: Device: PROCESS-INSTRUCTED SELF NEURO-MODULATION (PRISM)

INTERVENTIONS:
Device: PROCESS-INSTRUCTED SELF NEURO-MODULATION (PRISM) — Neurofeedback sessions targeting down-regulation of deep limbic structures, specifically the amygdala, delievered via PRISM: a non-significant risk device (software) intended to be used in research studies testing the clinical efficacy of an innovative paradigm for EEG-based neurofeedback.
  The study will include 12 EEG-NF sessions, administered twice per week for a duration of 6 "active" weeks in total. Twice weekly sessions will be held on non-consecutive days. Each session will last 30 minutes.
  EFP-EEG-NF training: Each NF training session consists of 5 consecutive sequences of NF presentations. During a "watch" condition (60 seconds) participants are instructed to passively view the animation, and are told that that the scenario does not influence their brain activity. In the "regulate" phase (60 seconds) participants are instructed to lower the room's unrest level. A "rest" phase (15 seconds) follows each sequence, allowing participants to relax.

SUMMARY:
This is a single-arm, open-label feasibility study. A maximum of 15 participants will be enrolled. All participants will undergo a novel neurofeedback intervention, targeting down-regulation of deep limbic structures, specifically the amygdalae. Participants will complete 12 neurofeedback sessions delivered twice weekly over 6 consecutive weeks. The intervention will be delivered via the PRISM platform.

ELIGIBILITY:
Inclusion Criteria:

* Adults ages 18-65 years
* Able to provide signed informed consent
* Any gender
* Diagnosis of PTSD as established by DSM-V
* 1 to 15 years since index trauma
* Taking a stable dose of SSRI antidepressants for at least 3 months OR un-medicated for at least 2 months
* Normal or corrected-to-normal vision
* Normal or corrected-to-normal hearing
* No intention of changing medication or psychotherapy for the duration of the study at the time of recruitment

Exclusion Criteria:

* Concurrent substance abuse
* Use of any prescribed benzodiazepine
* Lifetime bipolar disorder, psychotic disorder, autism, mental retardation. Comorbid mood and anxiety disorders will be permitted if they are not the primary focus of clinical attention
* Active suicidality within past year, or history of suicide attempt in past 2 years
* Any history of severe past drug dependence (i.e., a focus of clinical attention or a cause of substantial social or occupational difficulty)
* Any unstable medical or neurological condition
* Any history of brain surgery, of penetrating, neurovascular, infectious, or other major brain injury, of epilepsy, or of other major neurological abnormality (including a history of traumatic brain injury [TBI] with loss of consciousness for more than 24 hours or posttraumatic amnesia for more than 7 days)
* Any psychotropic medication other than a stable dose of selective serotonin reuptake inhibitors (SSRIs)
* Any change in accepted psychotropic medication within the past 2 months
* Recent initiation (within the past 3 months) of cognitive-behavioral therapy or any evidence-based PTSD psychotherapy (Cognitive Processing Therapy [CPT], Prolonged Exposure [PE], Eye Movement -Desensitization and Reprocessing [EMDR]); continuation of established maintenance supportive therapy will be permitted
* Significant hearing loss or severe sensory impairment
* Enrollment in another research study testing an experimental, clinical, or behavioral intervention intended to affect symptoms initiated within the last 2 months, or intended enrollment within the next 2.5 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-10-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
Change in CAPS-5 score from screening to completion | Screening visit (Week 0), and Post-Intervention Visit (Week 9)
  The CAPS-5 is a 30-item structured interview used to:
  * Make current (past month) diagnosis of PTSD
  * Make lifetime diagnosis of PTSD
  * Assess PTSD symptoms over the past week "1, 2" rule is used to determine a diagnosis: a frequency score of 1 (scale 0 = "none of the time" to 4 = "most or all of the time") and an intensity score 2 (scale 0 = "none" to 4 = "extreme") is required for a particular symptom to meet criterion.
  The assessor combines information about frequency and intensity of an item into a single severity rating. CAPS-5 total symptom severity score is calculated by summing severity scores for the 20 DSM-5 PTSD symptoms.
Change in PCL-5 score from baseline to completion | Baseline visit (Week 1), and Post-Intervention Visit (Week 9)
  The PCL-5 is a 20-item self-report measure that assesses the 20 DSM-5 symptoms of PTSD. The self-report rating scale is 0-4 for each symptom. A total symptom severity score (range - 0-80) can be obtained by summing the scores for each of the 20 items.

CONTACTS AND LOCATIONS:
Overall Officials: Charles Marmar, MD, Principal Investigator — NYU Langone Health
Locations (1):
- NYU Langone Health, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified participant data from the final research dataset used in the published manuscript will be shared upon reasonable request beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health. Requests may be directed to Lisa.Voltolina@nyulangone.org. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: beginning 9 months and ending 36 months following article publication or as required by a condition of awards and agreements supporting the research provided the investigator who proposes to use the data executes a data use agreement with NYU Langone Health.
Access Criteria: Requests may be directed to Lisa.Voltolina@nyulangone.org